CLINICAL TRIAL: NCT03634410
Title: SeniorWorkingLife (Danish Title: SeniorArbejdsLiv)
Acronym: SAL2018
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Research Centre for the Working Environment, Denmark (Other Government)
Collaborators: TrygFonden, Denmark (Industry); Team Arbejdsliv (Unknown); Aalborg University (Other); Statistics Denmark (Unknown)
Responsible Party: Principal Investigator, Lars L. Andersen, Professor, National Research Centre for the Working Environment, Denmark
Other Study IDs: 70103
Record Dates: First submitted 2018-08-10; First posted 2018-08-16 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Work Related Upper Limb Disorder; Musculoskeletal Pain; Work Accident; Work Injury; Work-Related Stress Disorder; Occupational Exposure; Occupation-related Stress Disorder
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Employed: people aged +50 and currently employed
- Unemployed: people aged +50 and currently unemployed
- Early retirement: people aged +50 and currently on early retirement
- Disability pension: people aged +50 and currently on disability pension

SUMMARY:
Due to demographic changes across Europe there are strong political interests in maintaining the labour force by prolonging working life, i.e. increasing retirement age. The present study investigates push and stay mechanisms for labor market attachment among older (+50 yrs) workers or people who have recently retired.

DETAILED DESCRIPTION:
Due to demographic changes across Europe there are strong political interests in maintaining the labour force by prolonging working life, i.e. increasing retirement age. The present study investigates push and stay mechanisms for labor market attachment among older workers or people who have recently retired. The study is a questionnaire survey, which is already funded. The ambition is to apply for further funding to do a cohort that is repeated every 2-3 years, as well as long-term register follow-up in Danish national registers about health and work.

The study has 4 target groups:

1. employed
2. unemployed
3. early retirement
4. disability pension

The questionnaire survey is sent to 30,000 Danish citizens and contains the following 14 areas:

1. Basic information (demographics, employment status etc.)
2. Broad overview of factors that may influence labor market attachment (health, working conditions, economic factors)
3. Role of the workplace
4. Age-discrimination
5. Economy
6. Specific questions about the possibility for 'early retirement' among employed and unemployed
7. Gradual retirement (e.g. possibility for reduced time or responsibility)
8. Competencies and continuing education/training of skills
9. Return-to-work
10. New technologies at the workplace
11. Job satisfaction and well-being
12. Working environment (physical, psychosocial etc.)
13. Lifestyle
14. Health and functional capacity

The study is supported by a grant from TrygFonden

ELIGIBILITY:
Inclusion Criteria:

Labor market status of:

* employed (employed at least 20/37 hours per week 1.quarter of 2018) OR
* unemployed (unemployed at least 20/37 hours per week 1.quarter of 2018) OR
* early retirement OR
* disability pension

Exclusion Criteria:

* those that do not fullfill the above inclusion criteria

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People in Denmark aged +50. The population will be drawn by Statistics Denmark
Sampling Method: Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychosocial Working Environment | Through study completion, an average of 2 year
  Psychosocial Working Environment is measured using questionnaire
Physical Working Environment | Through study completion, an average of 2 year
  Physical Working Environment is measured using questionnaire
Role of the workplace | Through study completion, an average of 2 year
  Role of the workplace is measured using questionnaire
Age-discrimination | Through study completion, an average of 2 year
  Age-discrimination is measured using questionnaire
Economy | Through study completion, an average of 2 year
  Economic status is measured using questionnaire
Early retirement | Through study completion, an average of 2 year
  Specific questions about the possibility for 'early retirement' among employed and unemployed
Gradual retirement | Through study completion, an average of 2 year
  Gradual retirement (e.g. possibility for reduced time or responsibility). Questionnaire
Competencies | Through study completion, an average of 2 year
  Competencies, education/training of skills will be evaluated using questionnaire
Return-to-work | Through study completion, an average of 2 year
  Possibilities for returning to work for those currently not employed will be evaluated using questionnaire
New technologies | Through study completion, an average of 2 year
  New technologies at the workplace will be evaluated using questionnaire
Job satisfaction | Through study completion, an average of 2 year
  Job satisfaction will be evaluated using questionnaire
Sickness absence | Through study completion, an average of 2 year
  Sickness absence will be evaluated through Danish registers
Disability pension | Through study completion, an average of 2 year
  Disability pension will be evaluated through Danish registers
Mortality | Through study completion, an average of 5 year
  Mortality will be evaluated through Danish registers

SECONDARY OUTCOMES:
Lifestyle | Through study completion, an average of 2 year
  Lifestyle will be evaluated using questionnaire
Health | Through study completion, an average of 2 year
  Health will be evaluated using questionnaire
Functional capacity | Through study completion, an average of 2 year
  Functional capacity will be evaluated using questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre for the Working Environment, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Due to the requirements for anonymity of participants in research projects in Denmark, it has not yet been decided how to share the data.
  People interested in performing analysis on the data should contact the research leader, Professor Lars L. Andersen, LLA@NRCWE.DK

REFERENCES:
- [Derived] Vinstrup J, Sundstrup E, Andersen LL. Psychosocial stress and musculoskeletal pain among senior workers from nine occupational groups: Cross-sectional findings from the SeniorWorkingLife study. BMJ Open. 2021 Mar 29;11(3):e043520. doi: 10.1136/bmjopen-2020-043520. PMID 33782021
- [Derived] Blafoss R, Skovlund SV, Lopez-Bueno R, Calatayud J, Sundstrup E, Andersen LL. Is hard physical work in the early working life associated with back pain later in life? A cross-sectional study among 5700 older workers. BMJ Open. 2020 Dec 7;10(12):e040158. doi: 10.1136/bmjopen-2020-040158. PMID 33293310
- [Derived] Skovlund SV, Blafoss R, Sundstrup E, Thomassen K, Andersen LL. Joint association of physical work demands and leg pain intensity for work limitations due to pain in senior workers: cross-sectional study. BMC Public Health. 2020 Nov 18;20(1):1741. doi: 10.1186/s12889-020-09860-6. PMID 33208134
- [Derived] Andersen LL, Sundstrup E. Study protocol for SeniorWorkingLife - push and stay mechanisms for labour market participation among older workers. BMC Public Health. 2019 Jan 31;19(1):133. doi: 10.1186/s12889-019-6461-6. PMID 30704447
- See also: SeniorArbejdsLiv — http://www.seniorarbejdsliv.dk/